CLINICAL TRIAL: NCT03234322
Title: A Cluster Randomized Trial to Investigate the Impact of a Type 2 Diabetes Risk Prediction Model on Change in Physical Activity Within Routine Health Checks in Primary Care.
Brief Title: The Impact of a Diabetes Risk Prediction Model in Primary Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Association of Statutory Health Insurance Physicians North Rhine (Unknown); German Institute of Human Nutrition (Other)
Responsible Party: Principal Investigator, Wolfgang Rathmann, PD Dr. Wolfgang Rathmann MSPH (USA), German Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DRT-Study
Record Dates: First submitted 2017-07-13; First posted 2017-07-31 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes Mellitus; Primary Prevention
Keywords: prevention; risk score; behaviour; physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: A pragmatic blinded parallel group superiority cluster randomized controlled trial. Clusters are PCPs (general practitioners, medical practitioners and internists working as general practitioners).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention group the routine health check is expanded by usage of a non-invasive diabetes risk score.
  Interventions: Other: external validated risk prediction model
- Control group (No Intervention): In the control group the routine health check is conducted.

INTERVENTIONS:
Other: external validated risk prediction model — The risk prediction model will be integrated into a routine health check. The diabetes risk prediction model contains modifiable non-invasive risk factors and consists of eleven questions on age, height, waist circumference, hypertension, physical activity, smoking status, intake of whole-grain bread, intake of red meat, coffee consumption, and family history of diabetes (parents and siblings) to predict the five-year diabetes risk. The filled diabetes risk score will be used in the counseling interview with the PCP at the end of the health check as a practical guide to discuss individual tailored preventive strategies.
  Other Names: The German Diabetes Risk Score
  Arms: Intervention group

SUMMARY:
Little evidence exists on the impact of diabetes risk scores, e.g. on physicians and patient's behavior, perceived risk of persons, shared-decision making and particularly on patient´s health. The aim of this study is to investigate the impact of a non-invasive diabetes risk prediction model in the primary health care setting as component of routine health checks on change in physical activity.

DETAILED DESCRIPTION:
Diabetes risk scores are predictive models to estimate the probability for an individual to develop diabetes within a defined time period. In the last years, many diabetes risk prediction models were developed worldwide. It has been proposed that using diabetes risk scores as first step of diabetes screening is more practical than blood glucose tests as the latter are time consuming and costly. Given the rapid development of diabetes risk scores and a simultaneous reluctance of primary care physicians (PCPs) to implement diabetes risk scores in everyday practice, there is an urgent need to expand our knowledge of the impact of diabetes risk scores in the primary health care setting. Thus, the aim of the study is to investigate the impact of a non-invasive risk prediction model in the primary health care setting as component of routine health checks on change in physical activity.

ELIGIBILITY:
Inclusion criteria for participation of medical practitioners:

* general practitioners, medical practitioners and internists working as general practitioners with and without further training in diabetology according to German Diabetes Association standards
* provide the routine health check

Exclusion criteria for participation of medical practitioners:

* treat exclusively patients with private insurance
* treat exclusively diabetes patients in a specialized medical practice

Inclusion criteria for participation of participants

* appointment for the routine health check
* insured in statutory health insurance
* age > 35 years
* Body Mass Index (BMI) of ≥ 27 kg/m2

Exclusion criteria for participation of participants

* type 1 or type 2 diabetes diagnosis or already abnormal blood glucose level (fasting glucose ≥ 126 mg/dl or 2 hours oral glucose tolerance test (oGTT) ≥ 200mg/dl or glycated hemoglobin (HbA1c) ≥6,5%) before the routine health check
* no sufficient German language skills to fill in the questionnaires
* presence of an incurable disease with a prognosis of less than one year
* severe mental illness or dementia
* severe underlying disease, which largely impairs physical activity
* pregnancy
* participation in another clinical study 30 days before study inclusion

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Difference of participant's physical activity at twelve months after the routine health check between the groups. | at baseline, 6 and 12 months follow-up
  Self-reported outcome, international validated questionnaire Physical Activity Questionnaire Short Last 7 Days Format (IPAQ-SF), which has been shown to be a reliable and valid tool to obtain comparable estimates of physical activity.

SECONDARY OUTCOMES:
Improvement in the counseling process assessed by PCPs. | at baseline and up to one year after the PCP entered the study
  Self-reported outcome, analyzed as difference in proportion of counseling regarding preventive strategies on balanced nutrition, body weight reduction, physical activity, and smoking secession between the groups. Questions are derived from a previous study.
Improvement in the counseling process assessed by participants. | at 6 months follow-up
  Self-reported outcome, analyzed as difference in proportion of counseling regarding preventive strategies on balanced nutrition, body weight reduction, physical activity, and smoking secession between the groups. Questions are derived from a previous study.
Improvement of shared decision making, assessed by participants. | at baseline
  Self-reported outcome, modified questionnaire to assess the difference in proportion of shared decision making for diabetes prevention opportunities between the groups.
Improvement of shared decision making, assessed by PCPs. | at baseline
  Self-reported outcome, modified questionnaire to assess the difference in proportion of shared decision making for diabetes prevention opportunities between the groups.
Improved motivation to change lifestyle, assessed by participants. | at baseline, 6 and 12 months follow-up
  Self-reported outcome, questions are based on the stage of change model to assess the stage of motivation according to weight reduction, physical activity, healthy diet, smoking cessation and were derived from previous studies. We will assess the difference of motivation change between the groups.
Change in Body-Mass-Index (BMI) | at baseline, 6 and 12 months follow-up
  At baseline, weight and height is objectively measured by the PCP, in the follow-up weight will be self-reported. We will analyse group differences in change of BMI at 6 and 12 months follow-up.
Change in participant's quality of life. | at baseline, 6 and 12 months follow-up
  Self-reported outcome, question has been derived from previous studies. We will assess the change of quality of life between the groups.
Change in participant's level of depression and anxiety. | at baseline, 6 and 12 months follow-up
  Self-reported outcomes, depression and anxiety will be assessed with a validated questionnaire, the Hospital Anxiety and Depression Scale (HADS-D). We will assess the change of depression and anxiety between the groups.
Change of participant's perceived risk of developing diabetes. | at baseline, 6 and 12 months follow-up
  Self-reported outcome by participants, questions derived from previous studies. We will assess the change in perceived risk between the groups.
Acceptance of PCPs according to the application of a diabetes risk score for routine use in clinical practice. | at baseline, and up to one year after the PCP entered the study
  Self-reported outcome, differences between the groups will be analyzed. Questions are derived from previous studies.
Acceptance of participants according to the application of a diabetes risk score for routine use in clinical practice. | at 6 months follow-up
  Self-reported outcome, questions derived from previous studies.

OTHER OUTCOMES:
Change on participant's individual diabetes risk. | at baseline, 6 and 12 months follow-up
  Self-reported outcome. Individual diabetes risk will be derived from the diabetes risk score in the intervention group at baseline, which is a validated questionnaire. In the follow-up questionnaires at 6 and 12 months, the questions of the diabetes risk score are included in the questionnaire of both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Rathmann, Prof., Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Institute for Biometrics and Epidemiology, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
Twelve months after data publication, de-identified data can be provided to other researchers upon request.
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: Universities and other non-profit organizations

REFERENCES:
- [Background] Dhippayom T, Chaiyakunapruk N, Krass I. How diabetes risk assessment tools are implemented in practice: a systematic review. Diabetes Res Clin Pract. 2014 Jun;104(3):329-42. doi: 10.1016/j.diabres.2014.01.008. Epub 2014 Jan 15. PMID 24485859
- [Background] Noble D, Mathur R, Dent T, Meads C, Greenhalgh T. Risk models and scores for type 2 diabetes: systematic review. BMJ. 2011 Nov 28;343:d7163. doi: 10.1136/bmj.d7163. PMID 22123912
- [Background] Godino JG, van Sluijs EM, Marteau TM, Sutton S, Sharp SJ, Griffin SJ. Lifestyle Advice Combined with Personalized Estimates of Genetic or Phenotypic Risk of Type 2 Diabetes, and Objectively Measured Physical Activity: A Randomized Controlled Trial. PLoS Med. 2016 Nov 29;13(11):e1002185. doi: 10.1371/journal.pmed.1002185. eCollection 2016 Nov. PMID 27898672
- [Background] Muller-Riemenschneider F, Holmberg C, Rieckmann N, Kliems H, Rufer V, Muller-Nordhorn J, Willich SN. Barriers to routine risk-score use for healthy primary care patients: survey and qualitative study. Arch Intern Med. 2010 Apr 26;170(8):719-24. doi: 10.1001/archinternmed.2010.66. PMID 20421559
- [Derived] Seidel-Jacobs E, Kohl F, Tamayo M, Rosenbauer J, Schulze MB, Kuss O, Rathmann W. Impact of applying a diabetes risk score in primary care on change in physical activity: a pragmatic cluster randomised trial. Acta Diabetol. 2022 Aug;59(8):1031-1040. doi: 10.1007/s00592-022-01895-y. Epub 2022 May 13. PMID 35551495
- [Derived] Jacobs E, Tamayo M, Rosenbauer J, Schulze MB, Kuss O, Rathmann W. Protocol of a cluster randomized trial to investigate the impact of a type 2 diabetes risk prediction model on change in physical activity in primary care. BMC Endocr Disord. 2018 Oct 16;18(1):72. doi: 10.1186/s12902-018-0299-2. PMID 30326888